CLINICAL TRIAL: NCT03432364
Title: A Phase 1/2, Open-label, Single-arm Study to Assess the Safety, Tolerability, and Efficacy of ST-400 Autologous Hematopoietic Stem Cell Transplant for Treatment of Transfusion-Dependent Beta-thalassemia (TDT)
Brief Title: A Study to Assess the Safety, Tolerability, and Efficacy of ST-400 for Treatment of Transfusion-Dependent Beta-thalassemia (TDT)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sangamo Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ST-400-01
Record Dates: First submitted 2018-02-01; First posted 2018-02-14 (Actual); Results first posted 2023-12-13 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-11

CONDITIONS: Transfusion Dependent Beta-thalassemia
Keywords: Beta thalassemia; Beta-thalassemia; Thalassemia major; Cooley's anemia; ZFN mediated genome editing; zinc finger nuclease
MeSH Terms: conditions — beta-Thalassemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ST-400 Investigational product (Experimental): ST-400 Investigational product is composed of autologous CD34+ hematopoietic stem/progenitor cells that are genetically modified ex vivo at the erythroid-specific enhancer of the BCL11A gene
  Interventions: Genetic: ST-400 Investigational product

INTERVENTIONS:
Genetic: ST-400 Investigational product — Single dose of ST-400 following chemotherapy conditioning with busulfan

SUMMARY:
This is a single-arm, multi-site, single-dose, Phase 1/2 study to assess ST-400 in 6 subjects with transfusion-dependent β-thalassemia (TDT) who are ≥18 and ≤40 years of age. ST-400 is a type of investigational therapy that consists of gene edited cells. ST-400 is composed of the patient's own blood stem cells which are genetically modified in the laboratory using Sangamo's zinc finger nuclease (ZFN) technology to disrupt a precise and specific sequence of the enhancer of the BCL11A gene (which normally suppresses fetal hemoglobin production in erythrocytes). This process is intended to boost fetal hemoglobin (HbF), which can substitute for reduced or absent adult (defective) hemoglobin. ST-400 is then infused back into the patient after receiving conditioning chemotherapy to make room for the new cells in the bone marrow, with the aim of producing new erythrocytes with increased amounts of HbF. The primary objective is to understand safety and tolerability of ST-400, and secondary objectives are to assess the effects on HbF levels and transfusion requirements.

DETAILED DESCRIPTION:
Once consented, study participants will progress through the following stages:

* Screening: in-person visit at the study site to confirm eligibility for proceeding
* Collection: autologous (self) blood stem cells are harvested at the study site, also known as apheresis
* Manufacturing of ST-400: no study participant activities expected
* Infusion: conditioning chemotherapy, followed by infusion of ST-400, occurs at the study site
* Follow-up: follow up at the study site to monitor for safety and effectiveness of the study

ELIGIBILITY:
Inclusion Criteria:

1. Informed Consent
2. Clinical diagnosis of TDT with ≥ 8 documented RBC transfusion events per year on an annualized basis in the 2-years prior to screening
3. Confirmed beta-thalassemia diagnosis by molecular genetic testing
4. Clinically stable and eligible to receive conditioning chemotherapy
5. Able and willing to use an effective method of contraception from the signing of the informed consent and for one year following ST-400 infusion.

Exclusion Criteria:

1. Previous history of autologous or allogeneic blood stem cell transplantation or solid organ transplantation
2. Pregnant or breastfeeding female
3. Medical contraindication to mobilization, apheresis, or conditioning
4. Significant liver, lung, heart, or kidney dysfunction
5. Diagnosis of HIV or evidence of active HBV or HCV
6. History of significant bleeding disorder or uncontrolled seizures
7. History of active malignancy in past 5 years (non-melanoma skin cancer or cervical cancer in situ permitted) any history of hematologic malignancy, or family history of cancer predisposition syndrome without negative testing result in the study candidate.
8. Currently participating in another clinical trial using an investigational study medication, or recent participation in such a trial
9. Previous treatment with gene therapy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2022-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sangamo Therapeutics, Inc.
Locations (6):
- United States (6):
  - University of California, Los Angeles, Los Angeles, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Dana-Farber Boston Children's Cancer and Blood Disorders Center, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brusson M, Miccio A. Genome editing approaches to beta-hemoglobinopathies. Prog Mol Biol Transl Sci. 2021;182:153-183. doi: 10.1016/bs.pmbts.2021.01.025. Epub 2021 Mar 1. PMID 34175041

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The original enrollment goal was six subjects were to be enrolled in the Phase 1/2 study ST-400-01, but 5 subjects were enrolled and dosed. One subject from the 5 dosed withdrew consent prior to completing the study. Subjects who received treatment with ST-400 were asked to participate in a separate observational long-term safety study.
Period: Primary (ST-400 Infusion up to Week 52 )
Arm/Group | ST-400 Investigational Product
Started | 5
Completed | 5
Not Completed | 0
Period: Follow Up (Weeks 52-156 Post Infusion)
Arm/Group | ST-400 Investigational Product
Started | 5
Completed | 4
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: The study population comprise male and non-pregnant, non-lactating female subjects with TDT between 18 and 40 years old, who are willing and able to undergo autologous HSCT.
Arm/Group | ST-400 Investigational Product
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.4 (7.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Sex: Female | 2
  Sex: Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5
Hemoglobin A (g/dL) at Baseline [Mean (Standard Deviation); unit: g/dL] | 11.040 (0.6006)
Hemoglobin F (g/dL) at Baseline [Mean (Standard Deviation); unit: g/dL] | 0.169 (0.0835)
Hemoglobin F Percentage at Baseline [Mean (Standard Deviation); unit: Percentage] | 1.48 (0.760)

OUTCOME MEASURES:

1. Primary Outcome: Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) up to 156 Weeks After the ST-400 Infusion
Description: Safety and tolerability assessed by number of participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) up to 156 weeks after the ST-400 infusion
Time Frame: Up to 156 weeks after the ST-400 infusion
Population: All subjects who received the ST-400 infusion
Measure: Number; unit: participants
Groups:
- ST-400 Investigational Product: ST-400 Investigational product is composed of autologous CD34+ hematopoietic stem/progenitor cells that are genetically modified ex vivo at the erythroid-specific enhancer of the BCL11A gene. Single dose of ST-400 following chemotherapy conditioning with busulfan.
Arm/Group | ST-400 Investigational Product
Number analyzed (Participants) | 5
participants
  Incidence of non-serious adverse events | 5
  Incidence of serious adverse events | 2

2. Secondary Outcome: Clinical Laboratory Measurement of Hemoglobin (Hb) Fractions (A and F in g/dL)
Description: Change from baseline clinical laboratory measurement of Hb fractions (A and F in g/dL) [Time Frame: Up to 156 weeks after ST-400 infusion]
Time Frame: Baseline, Weeks 26, 52, and 156 after ST-400 infusion
Population: Hb fractions (A and F in g/dL) Change from Baseline to Week 26, Week 52 and Week 156 in Safety Population
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | ST-400 Investigational Product
Number analyzed (Participants) | 5
g/dL
  Hemoglobin A (g/dL) Change from Baseline to Week 26 | -3.648 (2.0401)
  Hemoglobin A (g/dL) Change from Baseline to Week 52 | -3.227 (2.0789)
  Hemoglobin A (g/dL) Change from Baseline to Week 156 | -0.281 (1.5834)
  Hemoglobin F (g/dL) Change from Baseline to Week 26 | 1.025 (1.0898)
  Hemoglobin F (g/dL) Change from Baseline to Week 52 | 0.405 (0.2851)
  Hemoglobin F (g/dL) Change from Baseline to Week 156 | 0.502 (0.2936)

3. Secondary Outcome: Clinical Laboratory Measurements of Percent (%) HbF
Description: Change from baseline percent (%) HbF [Time Frame: Up to 156 weeks after ST-400 infusion]
Time Frame: Baseline, Weeks 26, 52, and 156 after ST-400 infusion
Population: Change Percent (%) HbF from Baseline to Week 26, Week 52 and Week 156 in Safety Population
Measure: Mean (Standard Deviation); unit: Percentage of Hemoglobin F
Arm/Group | ST-400 Investigational Product
Number analyzed (Participants) | 5
Percentage of Hemoglobin F
  Week 26 | 12.83 (14.282)
  Week 52 | 5.30 (3.188)
  Week 156 | 4.35 (3.040)

4. Secondary Outcome: Annualized Frequency of Packed RBC Transfusions
Description: Calculation of annualized frequency and volume of packed red blood cell (PRBC) transfusions after ST-400 infusion transfusion support in the 2 years prior to screening
Time Frame: From Baseline (2 years prior to screening/consent), to ST-400 Infusion (Day 0), after hematopoietic reconstitution and up to 156 weeks (post ST-400 infusion)
Population: Annualized Frequency of Blood Product Transfusion in Safety Population
Measure: Mean (Standard Deviation); unit: PRBC transfusions/year
Arm/Group | ST-400 Investigational Product
Number analyzed (Participants) | 5
PRBC transfusions/year
  Baseline transfusion support 2 years prior to screening/consent | 17.393 (5.4350)
  At ST-400 Infusion (Day 0) | 21.518 (4.8806)
  After hematopoietic reconstitution (up to 156 weeks after ST-400 infusion) | 19.665 (5.6716)

5. Secondary Outcome: Annualized Volume (mL) of Packed RBC Transfusions
Description: Historical baseline defined as transfusion support in the 2 years prior to screening.
Time Frame: as for outcome 4
Population: Blood Product Annualized Total Volume Transfused in Safety Population
Measure: Mean (Standard Deviation); unit: mL/year
Arm/Group | ST-400 Investigational Product
Number analyzed (Participants) | 5
mL/year
  Baseline transfusion support 2 years prior to screening/consent | 10295.984 (4063.3661)
  At ST-400 infusion (Day 0) | 7453.191 (4204.3456)
  After hematopoietic reconstitution (up to 156 weeks after ST-400 infusion) | 7068.788 (4480.8901)

ADVERSE EVENTS:
Time Frame: Participants with adverse events data collected from ICF signed through participant's last study visit, up to 156 weeks
Arm/Group | ST-400 Investigational Product
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 3/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ST-400 Investigational Product (N=5)
Drug withdrawal syndrome (General disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ST-400 Investigational Product (N=5)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4)
Anaemia (Blood and lymphatic system disorders) | 4 (8)
Neutropenia (Blood and lymphatic system disorders) | 3 (13)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (9)
Leukopenia (Blood and lymphatic system disorders) | 1 (8)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Tachycardia (Cardiac disorders) | 2 (4)
Palpitations (Cardiac disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (7)
Stomatitis (Gastrointestinal disorders) | 4 (8)
Diarrhoea (Gastrointestinal disorders) | 3 (5)
Nausea (Gastrointestinal disorders) | 5 (12)
Abdominal pain (Gastrointestinal disorders) | 1 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Haemoperitoneum (Gastrointestinal disorders) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 2 (5)
Bacterial sepsis (Infections and infestations) | 1 (1)
Coxsackie viral infection (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 5 (6)
Depression (Psychiatric disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Peripheral swelling (General disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (3)
Iron overload (Metabolism and nutrition disorders) | 2 (3)
Decreased appetite (Metabolism and nutrition disorders) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Fluid overload (Metabolism and nutrition disorders) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (5)
Hyperaesthesia (Nervous system disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 3 (5)
Road traffic accident (Injury, poisoning and procedural complications) | 2 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1)
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 (1)
Transfusion reaction (Injury, poisoning and procedural complications) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1)
Vaccination complication (Injury, poisoning and procedural complications) | 1 (2)
Platelet count decreased (Investigations) | 2 (10)
White blood cell count decreased (Investigations) | 2 (7)
Hepatic enzyme increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Bradypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Incision site pain (Injury, poisoning and procedural complications) | 1 (2)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Vascular access site pain (Injury, poisoning and procedural complications) | 3 (5)
International normalised ratio increased (Investigations) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Dysgeusia (Nervous system disorders) | 2 (3)
Haematuria (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to the limited sample size of 5 subjects, the study results presented are primarily descriptive in nature.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-04-09): https://cdn.clinicaltrials.gov/large-docs/64/NCT03432364/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-20): https://cdn.clinicaltrials.gov/large-docs/64/NCT03432364/SAP_001.pdf
  • Informed Consent Form (2020-05-14): https://cdn.clinicaltrials.gov/large-docs/64/NCT03432364/ICF_002.pdf